CLINICAL TRIAL: NCT03177499
Title: Virtual Imaging-based Early Portal Pressure Gradient (vePPG) After Placement of Transjugular Intrahepatic Portosystemic Shunts in Patients With Portal Hypertension
Brief Title: Virtual Imaging-based Early Portal Pressure Gradient (vePPG) (CHESS1702)
Acronym: vePPG
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Beijing Shijitan Hospital, Capital Medical University (Other); Beijing 302 Hospital (Other); The Third Xiangya Hospital of Central South University (Other); Xingtai People's Hospital (Other); Affiliated Traditional Chinese Medicine Hospital, Southwest Medical University (Unknown); First Affiliated Hospital, Sun Yat-Sen University (Other); Beijing Ditan Hospital (Other); PLA Army General Hospital (Unknown); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, M.D., Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHESS1702
Record Dates: First submitted 2017-06-04; First posted 2017-06-06 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Hypertension, Portal
Keywords: Portal pressure gradient; Transjugular intrahepatic portosystemic shunt; Virtual imaging-based portal pressure gradient
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Experimental): Patients will receive CT angiography, Doppler ultrasound, invasive PPG, and vePPG per protocol.
  Intervention: Procedure: Invasive PPG
  Interventions: Procedure: Invasive PPG

INTERVENTIONS:
Procedure: Invasive PPG — Invasive PPG obtained by means of catheterization.

SUMMARY:
Portal pressure gradient (PPG) above 12 mmHg after transjugular intrahepatic portosystemic shunt (TIPS) increases the risk of portal hypertension complications. Currently, a PPG reduction <12 mmHg after TIPS is the most consistent threshold associated with almost complete protection from variceal bleeding and ascites. However, the measurement of PPG requires an invasive procedure. A recent study investigated the variations in PPG measurements collected at different time points after placement of TIPS and demonstrated that a time point of at least 24 hours after which PPG values were best maintained (early PPG). It is of great clinical value to propose that an immediate PPG measurement fail to accurately identify the risk of decompensated event. And early PPG would change the decision making for re-intervention or not. However, the repeated invasive examination is extremely difficult to follow in clinical practice worldwide. The prospective multicenter trial aims to assess the diagnostic performance of a virtual imaging-based early portal pressure gradient (vePPG) (investigational technology) from CT angiography and Doppler ultrasound with invasive early PPG measurement as reference. The study participants with portal hypertension will be prospectively recruited at 10 high-volume liver centers in China.

DETAILED DESCRIPTION:
Portal pressure gradient (PPG) above 12 mmHg after transjugular intrahepatic portosystemic shunt (TIPS) increases the risk of portal hypertension complications. Currently, a PPG reduction <12 mmHg after TIPS is the most consistent threshold associated with almost complete protection from variceal bleeding and ascites. However, the measurement of PPG requires an invasive procedure. A recent study investigated the variations in PPG measurements collected at different time points after placement of TIPS and demonstrated that a time point of at least 24 hours after which PPG values were best maintained (early PPG). It is of great clinical value to propose that an immediate PPG measurement fail to accurately identify the risk of decompensated event. And early PPG would change the decision making for re-intervention or not. However, the repeated invasive examination is extremely difficult to follow in clinical practice worldwide. The prospective multicenter trial aims to assess the diagnostic performance of a virtual imaging-based early portal pressure gradient (vePPG) (investigational technology) from CT angiography and Doppler ultrasound with invasive early PPG measurement as reference. The study participants with portal hypertension will be prospectively recruited at 10 high-volume liver centers (Beijing Shijitan Hospital; 302 Hospital of PLA; Nanfang Hospital, Southern Medical University; The Third Xiangya Hospital of Central South University; Xingtai People's Hospital; Affiliated Traditional Chinese Medicine Hospital, Southwest Medical University; First Affiliated Hospital, Sun Yat-Sen University; Beijing Ditan Hospital; PLA Army General Hospital; Third Affiliated Hospital, Sun Yat-Sen University) in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients providing written informed consent
* Patients with portal hypertension and received the placement of TIPS
* Patients with invasive immediate PPG and early PPG measurement
* Has undergone > 64 multi-detector row CT angiography and Doppler ultrasound within 3 days prior to invasive early PPG measurement

Exclusion Criteria:

* Any severe adverse events after TIPS placement
* Inability to adhere to study procedures
* Prior devascularization operation
* Has received a liver transplant
* Patients with known anaphylactic allergy to iodinated contrast
* Pregnancy or unknown pregnancy status
* Patient requires an emergent procedure
* Any active, serious, life-threatening disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
vePPG Numerical Correlation | 1 day
  Correlation of vePPG numerical value with early PPG numerical value

SECONDARY OUTCOMES:
Immediate PPG Numerical Correlation | 7 days
  Correlation of immediate PPG numerical value with early PPG numerical value
Diagnostic Performance of vePPG | 1 day
  Accuracy, sensitivity, specificity, positive predictive value and negative predictive value of vePPG to determine re-intervention or not when compared to invasive early PPG as reference (PPG≥12mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Fuquan Liu, MD, Principal Investigator — Beijing Shijitan Hospital, Capital Medical University; Zhiwei Li, MD, Principal Investigator — Beijing 302 Hospital; Xiaolong Qi, MD, Study Chair — Nanfang Hospital, Southern Medical University
Locations (10):
- China (10):
  - 302 Hospital of PLA, Beijing, Beijing Municipality
  - Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - PLA Army General Hospital, Beijing, Beijing Municipality
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Xingtai People's Hospital, Xingtai, Hebei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Affiliated Traditional Chinese Medicine Hospital, Southwest Medical University, Luzhou, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garcia-Tsao G, Abraldes JG, Berzigotti A, Bosch J. Portal hypertensive bleeding in cirrhosis: Risk stratification, diagnosis, and management: 2016 practice guidance by the American Association for the study of liver diseases. Hepatology. 2017 Jan;65(1):310-335. doi: 10.1002/hep.28906. Epub 2016 Dec 1. No abstract available. PMID 27786365
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Silva-Junior G, Turon F, Baiges A, Cerda E, Garcia-Criado A, Blasi A, Torres F, Hernandez-Gea V, Bosch J, Garcia-Pagan JC. Timing Affects Measurement of Portal Pressure Gradient After Placement of Transjugular Intrahepatic Portosystemic Shunts in Patients With Portal Hypertension. Gastroenterology. 2017 May;152(6):1358-1365. doi: 10.1053/j.gastro.2017.01.011. Epub 2017 Jan 24. PMID 28130066
- [Background] Min JK, Leipsic J, Pencina MJ, Berman DS, Koo BK, van Mieghem C, Erglis A, Lin FY, Dunning AM, Apruzzese P, Budoff MJ, Cole JH, Jaffer FA, Leon MB, Malpeso J, Mancini GB, Park SJ, Schwartz RS, Shaw LJ, Mauri L. Diagnostic accuracy of fractional flow reserve from anatomic CT angiography. JAMA. 2012 Sep 26;308(12):1237-45. doi: 10.1001/2012.jama.11274. PMID 22922562
- [Background] Qi X, Li Z, Huang J, Zhu Y, Liu H, Zhou F, Liu C, Xiao C, Dong J, Zhao Y, Xu M, Xing S, Xu W, Yang C. Virtual portal pressure gradient from anatomic CT angiography. Gut. 2015 Jun;64(6):1004-5. doi: 10.1136/gutjnl-2014-308543. Epub 2014 Nov 14. No abstract available. PMID 25398771